CLINICAL TRIAL: NCT02271113
Title: A Randomized, Placebo Controlled, Phase1 Study to Assess the Safety and Pharmacokinetics of GMI-1271 in Healthy Adult Subjects
Brief Title: Phase I Study to Assess Safety and Pharmacokinetics of GMI-1271 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: GMI-1271-102
Record Dates: First submitted 2014-10-08; First posted 2014-10-22 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — uproleselan; enoxaparin sodium; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GMI-1271 (Experimental): IV GMI-1271
  Interventions: Drug: GMI-1271
- Placebo (Placebo Comparator): IV Placebo
  Interventions: Drug: Placebo
- Enoxaparin Sodium (Lovenox®) (Active Comparator): SC Lovenox®
  Interventions: Drug: Enoxaparin Sodium (Lovenox®)

INTERVENTIONS:
Drug: GMI-1271
  Arms: GMI-1271
Drug: Placebo
  Arms: Placebo
Drug: Enoxaparin Sodium (Lovenox®)
  Arms: Enoxaparin Sodium (Lovenox®)

SUMMARY:
In this study, the investigators will evaluate the safety, pharmacokinetics and effect on target biomarkers of coagulation, cell adhesion, and leukocyte and platelet activation of GMI-1271, an E-selectin antagonist, in healthy volunteers.

DETAILED DESCRIPTION:
Investigators will evaluate in a single ascending dose (SAD) and multiple ascending dose (MAD) fashion, the safety, pharmacokinetics and effect on target biomarkers of coagulation, cell adhesion, and leukocyte and platelet activation of GMI-1271, an E-selectin antagonist, in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Male or female
* Medically healthy, as defined by the absence of clinically significant screening results (e.g. laboratory profile, medical history, electrocardiogram (ECG), physical examination)
* BMI 18-35 kg/m2
* Voluntary consent to participate in the study
* No evidence of Lower Extremity Deep Vein Thrombosis (LE DVT) at baseline by ultrasound

Exclusion Criteria:

* Use of any prescription, investigational, herbal, supplemental, or over the counter medications including aspirin within 14 days (for the SAD phase) and 7 days (for the MAD phase) prior to day 1 or unwilling/unable to refrain from the use of these medications on days 1-8 for the SAD phase and days 1-12 of the MAD phase of the study
* Previous administration of GMI-1271
* Positive drug testing at screening and baseline or positive alcohol testing at baseline or unwilling/unable to refrain from the use of drugs or alcohol on days 1-8 for the SAD phase and days 1-12 for the MAD phase of the study
* Pregnant or breastfeeding
* Unwilling or unable to use contraception during the time of participation in the trial and 14 days afterwards (sexual abstinence is permissible)
* Positive HIV, Hepatitis B surface antigen or Hepatitis C antibody at screening
* Hypersensitivity or allergic reaction to compounds related to GMI-1271
* Use of moderate caffeine (≥ 300 mg/day) within 48 hours prior to dosing (day 1)
* History of bleeding disorder
* Any liver function test > 1.5 times upper limit of normal or renal insufficiency with creatinine clearance < 30 ml/min.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability | 14-19 days
  Adverse Event data review
Type of adverse events as a measure of safety and tolerability | 14-19 days
  Adverse Event data review
Severity of adverse events as a measure of safety and tolerability | 14-19 days
  Adverse Event data review
Review of lab results as a measure of Pharmacokinetics | 3-5 days
  Cmax (mg/mL)
Review of lab results as a measure of Pharmacokinetics | 3-5 days
  AUC (mg/mL)

SECONDARY OUTCOMES:
Incidence of bleeding | 14-19 days
  Adverse Event data review

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sood, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States